CLINICAL TRIAL: NCT03440736
Title: A Randomized, Multicenter 28 Week Study to Compare the Efficacy and Safety of Combining Cosentyx (Secukinumab) (4-weekly, 300 mg s.c.) With a Lifestyle Intervention to Cosentyx Therapy Alone in Adult Patients With Moderate to Severe Plaque-type Psoriasis and Concomitant Metabolic Syndrome, Followed by a 28 Week Extension Period
Brief Title: Comparison of Secukinumab 300 mg Combined With a Lifestyle Intervention to Secukinumab Alone for the Treatment of Moderate to Severe Psoriasis Patients With Concomitant Metabolic Syndrome
Acronym: METABOLYX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457ADE08; 2016-001671-79 (EudraCT Number)
Record Dates: First submitted 2018-01-31; First posted 2018-02-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Psoriasis; Metabolic Syndrome
Keywords: Psoriasis; Metabolic syndrome; Diabetes; Obesity; Life-style; Life-style intervention; Secukinumab; CAIN457A; CAIN457ADE08; AIN457A; Skin condition; skin disease; itching condition; psoriasis vulgaris; relapsing psoriasis; remitting psoriasis; immune-mediated systemic disease; skin lesions; red skin lesions; scaly patches; papules; plaques; itching
MeSH Terms: conditions — Psoriasis; Metabolic Syndrome; Diabetes Mellitus; Obesity; Skin Diseases; Plaque, Amyloid; Pruritus | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Secukinumab 300 mg subcutaneous (s.c.) (Active Comparator): Patients in arm A received therapy with Secukinumab 300 mg s.c., which consisted of two injections with 150 mg prefilled syringes at weeks 0, 1, 2, 3, 4, 8, 12, 16, 20 and 24 (last injection was performed at week 24).
  Interventions: Drug: Secukinumab
- Secukinumab 300 mg subcutaneous (s.c.) and lifestyle intervention (Experimental): Patients in arm B received therapy with Secukinumab 300 mg s.c., which consisted of two injections with 150 mg prefilled syringes at weeks 0, 1, 2, 3, 4, 8, 12, 16, 20 and 24 (last injection was performed at week 24). In addition they participated in a lifestyle intervention program.
  Interventions: Drug: Secukinumab; Behavioral: Life-style intervention

INTERVENTIONS:
Drug: Secukinumab — Secukinumab 300 mg s.c., which consisted of two injections with 150 mg prefilled syringes at weeks 0, 1, 2, 3, 4, 8, 12, 16, 20 and 24 (last injection was performed at week 24)
Behavioral: Life-style intervention — A structured program to guide weight loss and increased physical activity
  Arms: Secukinumab 300 mg subcutaneous (s.c.) and lifestyle intervention

SUMMARY:
This study was a randomized, open-label, parallel-group, active comparator controlled study with two treatment arms designed to answer the question whether the combination of Secukinumab with lifestyle intervention could primarily improve skin symptoms and secondly cardiometabolic status more than Secukinumab alone in psoriasis patients with concomitant metabolic syndrome by targeting the shared pathophysiology behind both diseases, which is systemic inflammation.

DETAILED DESCRIPTION:
This study included Core study with a duration of 28 weeks followed by an Extension period (exploratory period) with a duration of 28 weeks.

Core study:

After providing informed consent, patients were screened for eligibility for a period of 1 to 4 weeks prior to inclusion in the study. Eligible patients were randomized to one of the two treatment arms, which were the following:

* Arm A: Patients in arm A received a regular induction followed by 4-weekly maintenance treatment with secukinumab 300 mg s.c. until Week 28, where they completed the core study. The last secukinumab injection was to be administered at Week 24.
* Arm B: Patients in arm B received a regular induction followed by 4-weekly maintenance treatment with secukinumab 300 mg s.c. until Week 28. The last secukinumab injection was to be administered at Week 24. In addition to secukinumab treatment, patients in arm B participated in a lifestyle intervention program.

A biomarker sub-study was conducted during the core study in a subgroup of 100 patients (50 from each treatment arm).

The core study ended at Week 28.

Extension period (exploratory period):

After 28 weeks, the study continued with an extension period, during which lifestyle intervention was offered to all patients, irrespective of their prior treatment arm. This meant that patients of arm B, who were willing to, could continue their previously started lifestyle intervention program, and patients of arm A, who were willing to, could start the lifestyle intervention program at the beginning of the extension period. All patients, irrespective of their decision whether to start/continue lifestyle intervention or not, had to participate in the extension period and visit their dermatologic study center for scheduled visits. The extension period ended at Week 56, where all patients completed the study. No study drug was supplied during the extension period. The treating physician could choose psoriasis therapy freely according to their discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Men or women of at least 18 years of age at the time of screening.
3. Patients must be able to understand and communicate with the investigator and must be willing and able to comply with all study procedures.
4. Patients with moderate to severe plaque-type psoriasis who are candidates for systemic therapy, diagnosed at least 6 month before randomization and baseline value of

   * PASI > 10 and
   * DLQI > 10 and
   * Body Surface Area (BSA) affected by plaque-type psoriasis ≥ 10%
5. Fulfillment of Metabolic Syndrome definition (Alberti et al., 2009), which means fulfillment of ≥3 of the following criteria at screening visit:

   * Fasting (8 hours) plasma glucose ≥ 100 mg/dl or ongoing antidiabetic drug treatment (defined as: metformin, DPP4 inhibitors, GLP1 analogues, SGLT2 inhibitors)
   * Abdominal obesity defined by elevated waist circumference (measured as defined in section 6.4.5): Male: ≥94 cm, female: ≥80 cm (except for patients of Asian, South or Central American ethnicity, for whom the cut off values are: Male: ≥90 cm, female: ≥80 cm)
   * Fasting (8 hours) triglycerides ≥ 150 mg/dl or ongoing drug treatment for elevated triglycerides (defined as: fibrates or nicotinic acid).
   * Fasting (8 hours) HDL-C < 40 mg/dl in men or < 50 mg/dl in women or ongoing drug treatment for reduced HDL-C (defined as: fibrates, nicotinic acid or statins).
   * Resting blood pressure: Systolic blood pressure ≥ 130 and/ or diastolic blood pressure ≥ 85 mmHg (measured as defined in section 6.4.6) or ongoing antihypertensive drug treatment [defined as: ACE inhibitors, beta blockers, angiotensin receptor antagonists (e.g. Valsartan), aldosterone receptor antagonists, diuretics, nitrates, calcium channel blockers (e.g. Verapamil, Nifedipin), Aliskiren, Clonidin, alpha1 receptor antagonists (e.g. Doxazosin), Dihydralazin, Minoxidil, Moxonidin or Methyldopa].
6. Willingness and motivation to actively participate in a lifestyle intervention, which means patients need to be willing to increase physical activity and to change dietary habits.

Exclusion Criteria:

Patients fulfilling any of the following criteria are not eligible for inclusion in this study. No additional exclusions may be applied by the investigator, in order to ensure that the study population will be representative of all eligible patients.

1. Forms of psoriasis other than chronic plaque-type (e.g. pustular, erythrodermic and guttate psoriasis) at screening.
2. Previous exposure to Secukinumab or any other biologic drug directly targeting IL17A or the IL17A receptor (e.g. Brodalumab, Ixekizumab).
3. Exposure to anti-TNF treatment during 1 year prior to baseline.
4. Drug-induced psoriasis (i.e., new onset or current exacerbation from beta-blockers, calcium channel inhibitors or lithium) at screening.
5. History of hypersensitivity to Secukinumab, trehalose-dihydrate, L-histidine, L-histidinhydrochloride-monohydrate, L-methionine, polysorbate 80, water for injection, or to substances of similar chemical classes.
6. History of latex hypersensitivity.
7. Ongoing participation (including safety follow-up period) in other interventional or non-interventional studies in any dermatological indication
8. Ongoing use of prohibited treatments. Washout periods detailed in the protocol have to be adhered to (Table 5-1). Note: Administration of live vaccines 6 weeks prior to baseline (visit 2) or during the study period is also prohibited.
9. Diagnosis of type 1 diabetes.
10. Patients with diagnosed type 2 diabetes, if they fulfill one or more of the following conditions:

    * uncontrolled type 2 diabetes, meaning HbA1c > 8.0%,
    * pharmacological therapy with one or more of the following agents: Insulin, sulfonylurea agents/analogues, thiazolidinediones/glitazones
11. Insufficiently controlled, severe arterial hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 95 mmHg) with urgent need for therapy initiation or foreseeable need for medication change during the duration of the core study.
12. Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or within 30 days until the expected pharmacodynamic effect has returned to baseline, whichever is longer; or longer if required by local regulations.
13. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
14. Active ongoing inflammatory diseases other than psoriasis and psoriatic arthritis (PsA) that might confound the evaluation of the benefit of Secukinumab therapy.
15. Underlying conditions (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal) which in the opinion of the investigator significantly immunocompromises the subject and/or places the subject at unacceptable risk for receiving an immunomodulatory therapy.
16. Significant, progressive or uncontrolled medical problems at baseline which according to the opinion of the Investigator render the subject unsuitable for the trial - also in regard to participation in the lifestyle intervention - or put the subject at increased risk when participating in the trial (e.g. broken leg, congestive heart failure NYHA III/IV, uncontrolled hypertension with systolic ≥ 160 mmHg and/or diastolic ≥ 95 mmHg, severe uncontrolled asthma)
17. Medical history of myocardial infarction or angina pectoris
18. Any medical or psychiatric condition which, in the Investigator's opinion, would preclude the participant from adhering to the protocol or completing the study per protocol.
19. Serum creatinine level exceeding 2.0 mg/dl (176.8 μmol/L) at screening
20. Total white blood cell (WBC) count < 2,500/μl, or platelets < 100,000/μl or neutrophils < 1,500/μl or hemoglobin < 8.5 g/dl at screening.
21. Active systemic infections during the last two weeks (exception: common cold) prior to baseline (visit 2) or any infection that reoccurs on a regular basis.
22. History of an ongoing, chronic or recurrent infectious disease, or evidence of tuberculosis infection as defined by a positive QuantiFERON TB-Gold test (QFT) at screening. Subjects with a positive or indeterminate QFT test may participate in the study if full tuberculosis work up (according to local practice/guidelines) was completed within 12 weeks prior to visit 2 and establishes conclusively that the subject has no evidence of active tuberculosis. If presence of latent tuberculosis is established, then appropriate treatment must have been initiated at least 4 weeks prior to baseline (visit 2) and maintained according to local guidelines.
23. Past medical history record or current infection with HIV, hepatitis B or hepatitis C prior to baseline (visit 2).
24. History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system treated or untreated within the past 5 years, regardless of whether there is evidence of local recurrence or metastases (except for Bowen's disease, or basal cell carcinoma or actinic keratoses that have been treated with no evidence of recurrence in the past 12 weeks prior to baseline (visit 2); carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been removed).
25. Inability or unwillingness to undergo repeated venipuncture (e.g., because of poor tolerability or lack of access to veins).
26. History or evidence of ongoing alcohol or drug abuse, within the last six months before baseline (visit 2).
27. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using basic methods of contraception during dosing of investigational drug for at least 20 weeks after the end of Secukinumab treatment. Basic contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks before taking investigational drug. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 m prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject
    * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps).
    * Use of oral, (estrogen and progesterone), injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking investigational drug.
    * Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 781 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving Psoriasis Area and Severity Index (PASI) Score of 90 at week 28 | Baseline, Week 28
  The Psoriasis Area and Severity Index (PASI) is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, trunk, upper limbs, lower limbs); each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area * area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4).
  PASI 90 represents patients achieving >= 90% improvement (reduction) in PASI score compared to Baseline. Patients with missing PASI at Week 28 were counted as non-responders.

SECONDARY OUTCOMES:
Percentage of patients achieving Psoriasis Area and Severity Index (PASI) Score of 75 over time | Baseline, Week 1, Week 2, Week 3, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  The Psoriasis Area and Severity Index (PASI) is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, trunk, upper limbs, lower limbs); each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area * area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4).
  PASI 75 represents patients achieving >= 75% improvement (reduction) in PASI score compared to Baseline.
Percentage of patients achieving Psoriasis Area and Severity Index (PASI) Score of 90 over time | Baseline, Week 1, Week 2, Week 3, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  The Psoriasis Area and Severity Index (PASI) is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, trunk, upper limbs, lower limbs); each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area * area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4).
  PASI 90 represents patients achieving ≥ 90% improvement (reduction) in PASI score compared to Baseline.
Percentage of patients achieving Psoriasis Area and Severity Index (PASI) Score of 100 over time | Baseline, Week 1, Week 2, Week 3, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  The Psoriasis Area and Severity Index (PASI) is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, trunk, upper limbs, lower limbs); each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area * area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4).
  PASI 100 response/remission represents patients achieving complete clearing of psoriasis (PASI = 0) compared to Baseline.
Mean absolute Psoriasis Area and Severity Index (PASI) Score over time | Baseline, Week 1, Week 2, Week 3, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  The Psoriasis Area and Severity Index (PASI) is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, trunk, upper limbs, lower limbs); each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area * area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4).
  A negative change in absolute PASI score means that the severity of psoriasis has decreased, indicating an improvement in the patient's condition.
Mean change from Baseline in high-sensitivity C-reactive Protein (hsCRP) | Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  High-sensitivity C-reactive Protein (hsCRP) was evaluated in both treatment arms throughout the duration of the core study and summarized using descriptive statistics.
Mean change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 8, Week 16, Week 24, Week 28
  Hemoglobin A1c (HbA1c) was evaluated in both treatment arms throughout the duration of the core study and summarized using descriptive statistics.
Mean change from Baseline in Fructosamine | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  Fructosamine was evaluated in both treatment arms throughout the duration of the core study and summarized using descriptive statistics.
Mean change from Baseline in Fasting Plasma Glucose (FPG) | Baseline, Week 8, Week 16, Week 28
  Fasting Plasma Glucose (FPG) was evaluated in both treatment arms throughout the duration of the core study and summarized using descriptive statistics.
Mean change from Baseline in Total cholesterol | Baseline, Week 8, Week 16, Week 28
  Total cholesterol was evaluated in both treatment arms throughout the duration of the core study and summarized using descriptive statistics.
Mean change from Baseline in Low-Density Lipoprotein (LDL) | Baseline, Week 8, Week 16, Week 28
  Low-Density Lipoprotein (LDL) was evaluated in both treatment arms throughout the duration of the core study and summarized using descriptive statistics.
Mean change from Baseline in High-Density Lipoprotein (HDL) | Baseline, Week 8, Week 16, Week 28
  High-Density Lipoprotein (HDL) was evaluated in both treatment arms throughout the duration of the core study and summarized using descriptive statistics.
Mean change from Baseline in Triglycerides | Baseline, Week 8, Week 16, Week 28
  Triglycerides were evaluated in both treatment arms throughout the duration of the core study and summarized using descriptive statistics.
Mean change from Baseline in Waist circumference | Baseline, Week 1, Week 2, Week 3, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  Waist circumference was evaluated in both treatment arms throughout the duration of the core study and summarized using descriptive statistics.
Mean change from Baseline in Body weight | Baseline, Week 1, Week 2, Week 3, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  Body weight was evaluated in both treatment arms throughout the duration of the core study and summarized using descriptive statistics.
Mean change from Baseline in Body Mass Index (BMI) | Baseline, Week 1, Week 2, Week 3, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  Body Mass Index (BMI) was evaluated in both treatment arms throughout the duration of the core study and summarized using descriptive statistics.
Mean change from Baseline in Systolic Blood Pressure | Baseline, Week 1, Week 2, Week 3, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  Systolic Blood Pressure was evaluated in both treatment arms throughout the duration of the core study and summarized using descriptive statistics.
Mean change from Baseline in Diastolic Blood Pressure | Baseline, Week 1, Week 2, Week 3, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  Diastolic Blood Pressure was evaluated in both treatment arms throughout the duration of the core study and summarized using descriptive statistics.
Dermatology Life Quality Index (DLQI) Total Score over time | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  The Dermatology life Quality Index (DLQI) is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person. Each question refers to the impact of the skin disease on the patient's life (symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, treatment) over the previous week and is scored from 0 to 3, giving a possible score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).
Mean change from Baseline in Dermatology Life Quality Index (DLQI) Total Score over time | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  The Dermatology life Quality Index (DLQI) is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person. Each question refers to the impact of the skin disease on the patient's life (symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, treatment) over the previous week and is scored from 0 to 3, giving a possible score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).
Percentage of patients with Dermatology Life Quality Index (DLQI) Response | Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  All patients with DLQI score 0 and 1 were considered as responders and patients with DLQI score >=2 were considered as non-responders. Subjects with missing DLQI score were counted as non-responders.
World Health Organization Well-Being Index (WHO-5) Total score over time | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  The 5-item World Health Organization Well-Being Index (WHO-5) is a validated, short questionnaire consisting of 5 simple questions, assessing subjective psychological well-being of the respondents: Felt cheerful and in good spirits, Felt calm and relaxed, Felt active and vigorous, Feeling fresh and rested and Things that interest me in daily life. The recall period is the previous two weeks. Each item has 6 response categories, ranging from 5 ("the whole time") to 0 ("at no time point"). The raw score ranges from 0 to 25, with 0 representing worst possible and 25 representing best possible quality of life. To obtain a percentage score ranging from 0 to 100, the raw score is multiplied by 4. A percentage score of 0 represents worst possible, whereas a score of 100 represents best possible quality of life.
Mean change from Baseline in World Health Organization Well-Being Index (WHO-5) Total score over time | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  The 5-item World Health Organization Well-Being Index (WHO-5) is a validated, short questionnaire consisting of 5 simple questions, assessing subjective psychological well-being of the respondents: Felt cheerful and in good spirits, Felt calm and relaxed, Felt active and vigorous, Feeling fresh and rested and Things that interest me in daily life. The recall period is the previous two weeks. Each item has 6 response categories, ranging from 5 ("the whole time") to 0 ("at no time point"). The raw score ranges from 0 to 25, with 0 representing worst possible and 25 representing best possible quality of life. To obtain a percentage score ranging from 0 to 100, the raw score is multiplied by 4. A percentage score of 0 represents worst possible, whereas a score of 100 represents best possible quality of life.
Participant's self-assessed pain, itching and scaling over time | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  A self-administered, 11-point numeric rating scale (NRS, 0-10) was used to evaluate the subject's assessment of their current pain, itching and scaling. Respondents answered the following questions for the assessment of:
  * Pain: Overall, how severe was your psoriasis-related pain over the past 24 hours
  * Itching: Overall, how severe was your psoriasis-related itch over the past 24 hours
  * Scaling: Overall, how severe was your psoriasis-related scaling over the past 24 hours Subjects had to rate their pain, itching, and scaling from 0 to 10 (11-point scale), with the understanding that the 0 represented the absence or null end of the pain, itching, or scale intensity (i.e., no pain, itching or scaling) and the 10 represented the other extreme of pain, itching, or scaling intensity (i.e., pain, itching or scaling as bad as it could be). The number that the patient selected represented his or her intensity score.
Percentage change from Baseline in Participant's self-assessed pain, itching and scaling | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  A self-administered, 11-point numeric rating scale (NRS, 0-10) was used to evaluate the subject's assessment of their current pain, itching and scaling. Respondents answered the following questions for the assessment of:
  * Pain: Overall, how severe was your psoriasis-related pain over the past 24 hours
  * Itching: Overall, how severe was your psoriasis-related itch over the past 24 hours
  * Scaling: Overall, how severe was your psoriasis-related scaling over the past 24 hours Subjects had to rate their pain, itching, and scaling from 0 to 10 (11-point scale), with the understanding that the 0 represented the absence or null end of the pain, itching, or scale intensity (i.e., no pain, itching or scaling) and the 10 represented the other extreme of pain, itching, or scaling intensity (i.e., pain, itching or scaling as bad as it could be). The number that the patient selected represented his or her intensity score.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (57):
- Germany (57):
  - Novartis Investigative Site, Magdeburg, Sachen Anhalt
  - Novartis Investigative Site, Andernach
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Soden
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bramsche
  - Novartis Investigative Site, Braunschweig
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Detmold
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Falkensee
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Friedrichshafen
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Hagen
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanau
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Ibbenbueren
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Langenau
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lingen
  - Novartis Investigative Site, Löhne
  - Novartis Investigative Site, Lüdenscheid
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Memmingen
  - Novartis Investigative Site, Mönchengladbach
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Oberhausen
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Plauen
  - Novartis Investigative Site, Pommelsbrunn
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Quedlinburg
  - Novartis Investigative Site, Remscheid
  - Novartis Investigative Site, Seligenstadt
  - Novartis Investigative Site, Selters
  - Novartis Investigative Site, Simmern
  - Novartis Investigative Site, Soest
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Vechta
  - Novartis Investigative Site, Wuppertal

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

DOCUMENTS (2):
  • Study Protocol (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT03440736/Prot_002.pdf
  • Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT03440736/SAP_003.pdf